CLINICAL TRIAL: NCT01735175
Title: A Randomized, Double-blind, Parallel-group, Multi-center Phase 3 Comparative Study Investigating Efficacy and Safety of LA-EP2006 and Neulasta® in Breast Cancer Patients Treated With Myelosuppressive Chemotherapy
Brief Title: Phase III Study Comparing the Efficacy and Safety of LA-EP2006 and Neulasta®
Acronym: PROTECT-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Sandoz GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: LA-EP06-301; 2011-004532-58 (EudraCT Number)
Record Dates: First submitted 2012-11-22; First posted 2012-11-28 (Estimated); Results first posted 2017-06-15 (Actual); Last update posted 2017-08-07 (Actual); Status verified 2017-06

CONDITIONS: Neutropenic Complications; Breast Neoplasms; Chemotherapy-induced Neutropenia; Chemotherapeutic Toxicity
Keywords: biosimilars; Pegfilgrastim,; G-CSF,; neutropenia,; breast cancer,; myelosuppressive chemotherapy,; supportive care; granulocyte-colony-stimulating factor
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neulasta® (Active Comparator): During each chemotherapy cycle eligible patients receive Neulasta® s.c. post chemotherapy application.
  Interventions: Drug: Neulasta®
- LA-EP2006 (Experimental): During each chemotherapy cycle eligible patients receive LA-EP2006 s.c. post chemotherapy application.
  Interventions: Drug: LA-EP2006

INTERVENTIONS:
Drug: LA-EP2006 — Eligible patients are scheduled to receive six cycles of chemotherapy every three weeks. During each chemotherapy cycle pegfilgrastim is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim
  Arms: LA-EP2006
Drug: Neulasta® — Eligible patients are scheduled to receive six cycles of chemotherapy every three weeks. During each chemotherapy cycle pegfilgrastim is injected s.c. post chemotherapy application.
  Other Names: pegfilgrastim
  Arms: Neulasta®

SUMMARY:
The study will assess the efficacy of LA-EP2006 compared to Neulasta® with respect to the mean duration of severe neutropenia during treatment with myelosuppressive chemotherapy in breast cancer patients.

DETAILED DESCRIPTION:
This randomized, double-blind trial compared the proposed biosimilar LA-EP2006 with the reference Neulasta® in women (≥18 years) receiving chemotherapy for breast cancer. Therefore patients were randomized to receive LA-EP2006 (n = 159) or the reference product (n = 157) for ≤6 cycles of (neo)-adjuvant TAC (docetaxel 75mg/m^2, doxorubicin 50 mg/m^2, and cyclophosphamide 500mg/m^2) chemotherapy. The primary end point was the duration of severe neutropenia (DSN) during Cycle 1 (defined as number of consecutive days with absolute neutrophil count <0.5 × 10^9/l). The equivalence was confirmed if 95% CIs were within a ±1 day margin. LA-EP2006 was equivalent to the reference product in DSN (difference: 0.07 days; 95% CI [-0.12, 0.26]). Further, LA-EP2006 and the reference Neulasta® showed no clinically meaningful differences regarding efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven breast cancer
* eligible for six cycles of neoadjuvant or adjuvant chemotherapy

Exclusion Criteria:

* concurrent or prior chemotherapy for breast cancer
* concurrent or prior anti-cancer treatment for breast cancer such as endocrine therapy, immunotherapy, monoclonal antibodies, and/or biological therapy
* concurrent prophylactic antibiotics
* previous therapy with any G-CSF (granulocyte-colony stimulating factor) product

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Actual)
Dates: Start 2012-06; Primary Completion 2013-05 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Biopharmaceutical Clinical Development, Study Chair — Sandoz
Locations (37):
- Brazil (3):
  - Sandoz Investigational Site, Ijuí
  - Sandoz Investigational Site, Lajeado
  - Sandoz Investigational Site, Santo André
- India (6):
  - Sandoz Investigational Site, Andhra Pradesh
  - Sandoz Investigational Site, Delhi
  - Sandoz Investigational Site, Madurai
  - Sandoz Investigational Site, Maharashtra
  - Sandoz Investigational Site, Mumbai
  - Sandoz Investigational Site, Rajasthan
- Mexico (2):
  - Sandoz Investigational Site, Aguascalientes
  - Sandoz Investigational Site, Juchitán
- Romania (3):
  - Sandoz Investigational Site, Bucharest
  - Sandoz Investigational Site, Iași
  - Sandoz Investigational Site, Suceava
- Russia (14):
  - Sandoz Investigational Site, Barnaul
  - Sandoz Investigational Site, Bashkortostan
  - Sandoz Investigational Site, Berdsk
  - Sandoz Investigational Site, Ivanovo
  - Sandoz Investigational Site, Kabardino
  - Sandoz Investigational Site, Kazan'
  - Sandoz Investigational Site, Krasnodar
  - Sandoz Investigational Site, Kursk
  - Sandoz Investigational Site, Moscow
  - Sandoz Investigational Site, Oktyabrskaya
  - Sandoz Investigational Site, Ryazan
  - Sandoz Investigational Site, Saint Petersburg
  - Sandoz Investigational Site, Tula
  - Sandoz Investigational Site, Veliky Novgorod
- Ukraine (9):
  - Sandoz Investigational Site, Cherkasy
  - Sandoz Investigational Site, Chernivtsi
  - Sandoz Investigational Site, Dnipropetrovsk
  - Sandoz Investigational Site, Kharkiv
  - Sandoz Investigational Site, Kryvyi Rih
  - Sandoz Investigational Site, Luhansk
  - Sandoz Investigational Site, Mariupol
  - Sandoz Investigational Site, Vinnytsia
  - Sandoz Investigational Site, Zaporizhzhia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Harbeck N, Lipatov O, Frolova M, Udovitsa D, Topuzov E, Ganea-Motan DE, Nakov R, Singh P, Rudy A, Blackwell K. Randomized, double-blind study comparing proposed biosimilar LA-EP2006 with reference pegfilgrastim in breast cancer. Future Oncol. 2016 Jun;12(11):1359-67. doi: 10.2217/fon-2016-0016. Epub 2016 Mar 29. PMID 27020170
- [Derived] Blackwell K, Gascon P, Jones CM, Nixon A, Krendyukov A, Nakov R, Li Y, Harbeck N. Pooled analysis of two randomized, double-blind trials comparing proposed biosimilar LA-EP2006 with reference pegfilgrastim in breast cancer. Ann Oncol. 2017 Sep 1;28(9):2272-2277. doi: 10.1093/annonc/mdx303. PMID 28637287

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LA-EP2006 | Neulasta®
Started (Allocated) | 159 | 157
Completed All Cycles | 141 | 150
Completed All Treatments as Planned | 140 | 150
Completed the 6-month SFU Visit (1 more patient, LA-EP06 arm died due to disease progression, not included in participant flow-death) | 120 | 138
Completed (Completed the study as planned (prior to Safety follow-up)) | 130 | 144
Not Completed | 29 | 13
Not completed — Withdrawal by Subject | 9 | 2
Not completed — Lost to Follow-up | 4 | 2
Not completed — Death | 3 | 2
Not completed — Other (mostly EOS/EOT visit missing) | 13 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LA-EP2006 | Neulasta® | Total
Number analyzed (Participants) | 159 | 157 | 316
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.9 (9.53) | 50.5 (10.87) | 50.2 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 157 | 316
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 18 | 29
  Not Hispanic or Latino | 148 | 139 | 287
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — More than one race patients (n = 6) were of Mestizo or Parda origin.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 28 | 26 | 54
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 0 | 0
    White | 129 | 127 | 256
    More than one race | 2 | 4 | 6
    Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI is missing for 1 patient allocated to Neulasta®
  kg/m^2
    number analyzed (Participants) | 159 | 156 | 315
    (all) | 27.47 (26.76) | 27.44 (26.35) | 27.45 (26.40)
Time since diagnosis [Median (Full Range); unit: months] — For 4 patients in the LA-EP2006 treatment group, time since initial diagnosis was > 12 months. It was confirmed by the respective study site that the patients had not received treatment between diagnosis and study entry. Population: For 6 patients in the LA-EP2006 treatment group and 10 patients in the Neulasta® treatment group, the date of initial diagnosis was incomplete.
  months
    number analyzed (Participants) | 153 | 147 | 300
    (all) | 1.35 [0.1 to 76.0] | 1.38 [0.2 to 10.9] | 1.38 [0.1 to 76.0]
Disease stage [Count of Participants; unit: Participants] — TNM Disease stage was defined according to the American Joint Committee on Cancer (AJCC): (I) = T1 N0 M0 / T0 N1mi M0 / T1 N1mi M0; (II) = T0 N1 M0 / T1 N1 M0 / T2 N0 M0 / T2 N1 M0 / T3 N0 M0; (III) = T0 N2 M0 / T1 N2 M0 / T2 N2 M0 / T3 N1 M0 / T3 N2 M0 / T4 N0 M0 / T4 N1 M0 / T4 N2 M0 / AnyT N3 M0; (IV) = AnyT AnyN M1; T: size or direct extent of the primary tumour; N: degree of spread to regional lymph nodes; N1mi: Micrometastases (> 0.2 mm and/or > 200 cells, but none > 2.0 mm); M: presence of distant; https://www.cancer.gov/types/breast/hp/breast-treatment-pdq#link/_27
  Participants
    I | 4 | 3 | 7
    II | 74 | 73 | 147
    III | 81 | 78 | 159
    IV | 0 | 3 | 3
Previous breast cancer surgery [Count of Participants; unit: Participants] | 149 | 146 | 295
Previous radiotherapy [Count of Participants; unit: Participants] | 7 | 9 | 16
ECOG performance status [Count of Participants; unit: Participants] — ECOG = Eastern Cooperative Oncology Group
  Participants
    0 (fully active) | 128 | 123 | 251
    1 (restricted in physically strenuous activity) | 31 | 34 | 65

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Severe Neutropenia (DSN) During Cycle 1 of Chemotherapy
Description: Mean duration of severe neutropenia, defined as number of consecutive days with ANC <0.5 × 10^9 cells/L (grade 4 neutropenia).
Time Frame: 21 days (Cycle 1 of chemotherapy treatment)
Population: FAS set = full analysis set; PP set = per protocol set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
days
  FAS: number analyzed (Participants) | 155 | 155
  FAS | 0.75 (0.878) | 0.83 (0.898)
  PP: number analyzed (Participants) | 146 | 149
  PP | 0.75 (0.875) | 0.79 (0.872)
Statistical Analysis 1: Comparison: LA-EP2006 vs Neulasta®; The hierarchical test procedure aimed to show that 1. LA-EP2006 and Neulasta® are equivalent with respect to DSN duration in Cycle 1 (margin±1 day), and, if so 2. LA-EP2006 is non-inferior to Neulasta® with respect to DSN duration in Cycle 1 (margin of -0.6 days); Test type: Equivalence — The testing procedure was set up in a hierarchical structure, where first equivalence between LA-EP2006 and Neulasta® was assessed (margin ±1 day) and only if this was successfully established, non-inferiority between the two products was tested using a tighter margin of -0.6 days; p = 0.05, ANCOVA; The primary endpoints was analyzed with analysis of covariance (ANCOVA); Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.12 to 0.26] — The difference between LA-EP2006 and reference pegfilgrastim was 0.07 days (95% CI [-0.12, 0.26]). 95% CIs were within the predefined margin of ±1 day confirming equivalence
Statistical Analysis 2: Comparison: LA-EP2006 vs Neulasta®; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — The testing procedure was set up in a hierarchical structure, where first equivalence between LA-EP2006 and Neulasta was assessed (margin ±1 day) and only if this was successfully established, non-inferiority between the two products was tested using a tighter margin of -0.6 days; p = 0.05, ANCOVA; The primary endpoints was analyzed with analysis of covariance (ANCOVA); Mean Difference (Net) = 0.07, 95% CI 2-sided [-0.12 to 0.26] — LA-EP2006 is non-inferior to Neulasta® because the lower bound of the 95% CI is entirely above the non-inferiority margin of -0.6 days

2. Secondary Outcome: Incidence of Febrile Neutropenia (FN)
Description: FN was defined as an oral temperature ≥ 38.3°C while having an absolute neutrophil count (ANC) < 0.5 × 10^9 cells/L. Serious treatment-emergent adverse events (TEAEs) were reconciled with the fever and ANC results recorded in the patient diary and CRF and therefore only the serious TEAEs of FN ("febrile neutropenia", "neutropenic sepsis") were taken into account.
Time Frame: across all cycles (18 weeks)
Population: Number of patients with at least one episode of febrile neutropenia by cycle and across all cycles (FAS set)
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
Participants
  Cycle 1 | 6 | 11
  Cycle 2 | 2 | 1
  Cycle 3 | 2 | 1
  Cycle 4 | 1 | 0
  Cycle 5 | 2 | 0
  Cycle 6 | 1 | 1
  All cycles (at least on incidence) | 9 | 12

3. Secondary Outcome: Number of Patients With at Least One Episode of Fever by Cycle and Across All Cycles
Description: Fever was defined as an oral temperature ≥ 38.3°C. Fever episodes were characterized by maximum oral temperature and the number of patients who had fever at least once.
Time Frame: across al cycles (18 weeks)
Population: Patients with more than 1 event during the study (overall) are counted only once. FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
Participants
  Cycle 1 | 9 | 14
  Cycle 2 | 6 | 2
  Cycle 3 | 7 | 6
  Cycle 4 | 5 | 2
  Cycle 5 | 7 | 4
  Cycle 6 | 5 | 3
  Overall | 26 | 26

4. Secondary Outcome: Depth of ANC Nadir in Cycle 1
Description: The depth of ANC nadir was defined as the patient's lowest ANC (10^9 cells/L) in Cycle 1. Only the evaluable patients with a depth of ANC in Cycle 1 are given.
Time Frame: Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 156 | 155
10^9 cells/L | 1.102 (1.5398) | 0.921 (1.1771)

5. Secondary Outcome: Number of Patients With ANC Nadir Per Day in Cycle 1
Description: Numbers of patients with ANC nadir based per day during Cycle 1 are given.
Time Frame: Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
Participants
  Days 1-5 | 5 | 5
  Day 6 | 7 | 4
  Day 7 | 101 | 104
  Day 8 | 34 | 25
  Day 9 | 1 | 7
  Days 10-15 | 8 | 10

6. Secondary Outcome: Time to ANC Recovery in Days in Cycle 1
Description: Time to absolute neutrophil count (ANC) recovery in Cycle 1 was defined as the time in days from ANC nadir until the patient's ANC had increased to ≥ 2 × 10^9 cells/L. Only the evaluable patients with a depth of ANC in Cycle 1 and a later increase of ANC ≥ 2 × 10^9 cells/L are given.
Time Frame: across Cycle 1 (3 weeks)
Population: FAS set = full analysis set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 154 | 154
days | 1.58 (1.053) | 1.72 (1.100)

7. Secondary Outcome: Frequency of Infections by Cycle and Across All Cycles
Description: The number of patients with infections was recorded for each cycle and across all cycles. Infections were identified by the AE documentation page selecting all events coded with System Organ Class "Infections and Infestations".
Time Frame: across all cycles (18 weeks)
Population: Patients with more than 1 event during the study (overall) are counted only once. FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
Participants
  Cycle 1 | 7 | 4
  Cycle 2 | 6 | 5
  Cycle 3 | 3 | 8
  Cycle 4 | 2 | 3
  Cycle 5 | 11 | 4
  Cycle 6 | 5 | 3
  Overall | 22 | 24

8. Secondary Outcome: Mortality Due to Infection
Description: Number of patients with death due to infections
Time Frame: Study course (41 weeks)
Population: FAS set = full analysis set
Measure: Count of Participants; unit: Participants
Arm/Group | LA-EP2006 | Neulasta®
Number analyzed (Participants) | 159 | 157
Participants
  Yes | 0 | 2
  No | 159 | 155

ADVERSE EVENTS:
Time Frame: Patients were followed for a 6-month safety period from the last administration of pegfilgrastim.
Description: If not otherwise specified, only treatment-emergent adverse event (TEAEs) (i.e. AEs with a date of onset on or after the date of the first administration of chemotherapy and not later than 30 days after the last dose of chemotherapy) and post-TEAEs (i.e. AEs with a date of onset after the time point of 30 days after the last chemotherapy administration) are reported. SAF set = safety analysis set was used
Arm/Group | LA-EP2006 | Neulasta®
All-Cause Mortality (participants affected / at risk) | 4/159 | 2/157
Serious Adverse Events (participants affected / at risk) | 16/159 | 21/157
Other Adverse Events (participants affected / at risk) | 140/159 | 128/157
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LA-EP2006 (N=159) | Neulasta® (N=157)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 12
Neutropenia (Blood and lymphatic system disorders) | 3 | 6
Anemia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 2 | 0
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Asthenia (General disorders) | 1 | 0
Disease progression (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Thrombophlebitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Delirium febrile (Psychiatric disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LA-EP2006 (N=159) | Neulasta® (N=157)
Neutropenia (Blood and lymphatic system disorders) | 25 | 30
Vascular disorders (Vascular disorders) | 9 | 10
Cardiac disorders (Cardiac disorders) | 1 | 5
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 82 | 79
Erythema (Skin and subcutaneous tissue disorders) | 14 | 16
Asthenia (General disorders) | 63 | 56
Fatigue (General disorders) | 18 | 21
Pyrexia (General disorders) | 9 | 12
Pain (General disorders) | 7 | 10
Odema peripheral (General disorders) | 10 | 5
Nausea (Gastrointestinal disorders) | 64 | 58
Vomitting (Gastrointestinal disorders) | 34 | 32
Diarrhoe (Gastrointestinal disorders) | 23 | 31
Stomatitis (Gastrointestinal disorders) | 8 | 13
Constipation (Gastrointestinal disorders) | 10 | 9
Abdominal pain (Gastrointestinal disorders) | 8 | 7
Anemia (Blood and lymphatic system disorders) | 16 | 17
Leukopenia (Blood and lymphatic system disorders) | 11 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 7 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Respiratory tract infection viral (Infections and infestations) | 3 | 9
Respiratory tract infection (Infections and infestations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 8
Headache (Nervous system disorders) | 5 | 9
Alanine aminotransferase increased (Investigations) | 6 | 3
Aspatate aminotransferase increased (Investigations) | 6 | 2
Weight decreased (Investigations) | 3 | 5
Gamma-glutamyltransferase increased (Investigations) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes